CLINICAL TRIAL: NCT01692587
Title: Does Protein Restriction Inhibit Prostrate Cancer Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201011804
Record Dates: First submitted 2012-09-07; First posted 2012-09-25 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
Keywords: PSA; protein; prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No changes in dietary group
- Protein restrictive diet (Experimental): reduced protein diet
  Interventions: Other: Protein restrictive diet

INTERVENTIONS:
Other: Protein restrictive diet — To begin a reduced protein diet
  Arms: Protein restrictive diet

SUMMARY:
The Purpose of the Protein Study is to investigate whether a reduced protein diet can inhibit the growth of prostate cancer in humans.

The Investigators hypothesis is that a reduced protein diet will inhibit expression of genes that are involved in the growth of prostate cancer.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether or not a low protein diet has an inhibitory effect on prostate cancer cell growth.

The primary outcome measures relative to the investigators primary objectives are:

For Group 1 the expression of genes and proteins of the PI-3K/Akt/mTOR pathway. For Group 2 the PSA values obtained every three months.

ELIGIBILITY:
Inclusion Criteria:

group 1

1. Patient must have a diagnosis of prostate cancer confirmed by pathology.
2. Patient must be scheduled to undergo radical prostatectomy no sooner than 6 weeks from date of enrollment (to allow for a minimum of 4 weeks on the low protein diet).
3. Patient must have adequate baseline protein intake (screening 4-day food record shows protein > 1.0 g/kg FFM)
4. Patient must be able to understand the English-language instructions.
5. Patient must be able to comply with the low protein diet (as evaluated by the dietitian and other study team members).
6. Patient must be able to understand and willing to sign an IRB-approved written informed consent document.

5.2.2 Inclusion Criteria - Group 2

1. Patient must have a diagnosis of prostate cancer.
2. Patient must have previously undergone a radical prostatectomy for treatment of prostate cancer.
3. Patient must have a detectable PSA (defined as PSA ≥ 0.1) in at least two consecutive measurements, taken at least one month apart, with no therapy between the PSA measurements. If the patient has had additional therapy after the radical prostatectomy, there must be evidence of a rising PSA (i.e., two consecutive measurements at least one month apart) after the patient has completed the intervening therapy (meaning that the patient must have failed treatment).
4. Patient must have adequate baseline protein intake (screening 4-day food record shows protein > 1.0 g/kg FFM).
5. Patient must have adequate baseline caloric intake (screening 4-day food record shows caloric intake of > 1500 kcal/day).
6. Patient must be able to understand the English-language instructions.
7. Patient must be able to comply with the low protein diet (as evaluated by the dietitian and other study team members).
8. Patient must be able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

1. Patient must not currently be receiving any therapy for prostate cancer.
2. Patient must not have any serious chronic illness such as unstable angina, any uncontrolled metabolic disorder, or any immunologic disorder.
3. Patient must not have a history of any previous malignancy (with the exception of squamous or basal cell carcinoma of the skin) in the 5 years prior to enrollment (for Group 1) or 12 months prior to enrollment (for Group 2).
4. Patient must not have a previous history of a stroke.
5. Patient must not be taking any medications that might confound the study results (anabolic agents (such as androgen, androgen precursor, rhGH) in the 6 months prior to enrollment; corticosteroids (other than nasal) in the 6 months prior to enrollment; or finasteride or dutasteride).
6. Patient must not have dementia or any other cognitive impairment.
7. Patient must not have a lifestyle or fixed diet pattern that would interfere with participation in or interpretation of the results of this study

   -

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Group1--Expression of genes and proteins of the PI-3K/Akt/mTOR pathway. Group 2--PSA values obtained every three months | group 1- (4-6 weeks), group 2 -(52 weeks)
  The investigators will be looking at the increase or decrease of PSA values between control and protein restricted diet participants obtained for the length of study.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Fontana, MD,PhD, Principal Investigator — Washington University School of Medicine; Valeria Tosti, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Plan to publish

REFERENCES:
- [Background] Fontana L, Cummings NE, Arriola Apelo SI, Neuman JC, Kasza I, Schmidt BA, Cava E, Spelta F, Tosti V, Syed FA, Baar EL, Veronese N, Cottrell SE, Fenske RJ, Bertozzi B, Brar HK, Pietka T, Bullock AD, Figenshau RS, Andriole GL, Merrins MJ, Alexander CM, Kimple ME, Lamming DW. Decreased Consumption of Branched-Chain Amino Acids Improves Metabolic Health. Cell Rep. 2016 Jul 12;16(2):520-530. doi: 10.1016/j.celrep.2016.05.092. Epub 2016 Jun 23. PMID 27346343
- [Background] Trevino-Villarreal JH, Reynolds JS, Bartelt A, Langston PK, MacArthur MR, Arduini A, Tosti V, Veronese N, Bertozzi B, Brace LE, Mejia P, Trocha K, Kajitani GS, Longchamp A, Harputlugil E, Gathungu R, Bird SS, Bullock AD, Figenshau RS, Andriole GL, Thompson A, Heeren J, Ozaki CK, Kristal BS, Fontana L, Mitchell JR. Dietary protein restriction reduces circulating VLDL triglyceride levels via CREBH-APOA5-dependent and -independent mechanisms. JCI Insight. 2018 Nov 2;3(21):e99470. doi: 10.1172/jci.insight.99470. PMID 30385734
- [Background] Eitan E, Tosti V, Suire CN, Cava E, Berkowitz S, Bertozzi B, Raefsky SM, Veronese N, Spangler R, Spelta F, Mustapic M, Kapogiannis D, Mattson MP, Fontana L. In a randomized trial in prostate cancer patients, dietary protein restriction modifies markers of leptin and insulin signaling in plasma extracellular vesicles. Aging Cell. 2017 Dec;16(6):1430-1433. doi: 10.1111/acel.12657. Epub 2017 Sep 17. PMID 28921841